CLINICAL TRIAL: NCT06014944
Title: A Single-arm, Single-center, Prospective Clinical Study of Short-course Radiotherapy Combined With Furoquintinib and PD-1 Monoclonal Antibody for Neoadjuvant Therapy of PMMR/MSS Type Middle and Low Locally Advanced Rectal Cancer
Brief Title: Short-course Radiotherapy Combined With Furoquintinib and PD-1 Monoclonal Antibody
Acronym: PMMR/MSS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhang, Director of the department of colorectal surgery, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHoicelll
Record Dates: First submitted 2023-07-28; First posted 2023-08-28 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Rectal Cancer
Keywords: short course radiotherapy; furoquintinib; PD-1; low locally advanced rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short-course radiotherapy combined with furoquintinib and PD-1 monoclonal antibody (Experimental): Radiotherapy 5 * 5 Gy, once a day, 5 Gy each time, for 5 days.Two weeks after the end of radiotherapy, the patients were treated with furoquintinib combined with slurimab, furoquintinib 5 mg / time / day, d1-14, Q3 W ; combined with 300 mg of brucella, intravenous injection, d1, Q3W ; a total of 4 cycles of treatment.
  Interventions: Drug: Short-course radiotherapy combined with furoquintinib and PD-1 monoclonal antibody

INTERVENTIONS:
Drug: Short-course radiotherapy combined with furoquintinib and PD-1 monoclonal antibody — neoadjuvant therapy for short-course radiotherapy combined with furoquintinib and PD-1 monoclonal antibody for PMMR / MSS type middle and low locally advanced rectal cancer.

SUMMARY:
The investigators conduct a single-arm, single-center, prospective clinical study enrolling patients diagnoses with pMMR / MSS type middle and low locally advanced rectal cancer who had not received systemic anti-tumor therapy to explore the efficacy and safety of short-course radiotherapy combined with furoquintinib and PD-1 monoclonal antibody as neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. This study has been fully understood and voluntarily signed informed consent ;
2. Age 18-75 years old ( including 18 and 75 years old ) ; rectal adenocarcinoma was histologically confirmed as pMMR / MSS type ( according to the detection criteria of the institutional testing center, it can be detected by immunohistochemistry, PCR or NGS ), and was staged as stage II ( T3-4N0 ) or stage III ( T1-4N1-2 ) by MRI and CT.

4.MRI was used to evaluate the middle and low rectal cancer below 10 cm from the anal margin of the tumor ; 5.Patients who were recommended for neoadjuvant therapy after evaluation by the Multidisciplinary Oncology Committee ; 6.ECOG physical condition 0-1 points ; 7.Expected survival ≥ 2 years ; 8.No previous anti-tumor treatment has been received ; the function of vital organs meets the following requirements ( not allowed to use any blood components and cell growth factors within * 14 days before enrollment ) : Absolute neutrophil count ≥ 1.5 × 109 / L ; platelet ≥ 100 × 109 / L ; hemoglobin ≥ 90g / L ; total bilirubin < 1.5 times ULN ; aLT and / or AST < 2.5 times ULN ; serum creatinine < 1.5 times ULN ; endogenous creatinine clearance rate ≥ 50ml / min ; 10. Women of childbearing age need to take effective contraceptive measures ; 11.good compliance, with follow-up.

Exclusion Criteria:

* 1.Unable to comply with the research program or research procedures ; 2.Patients with surgical taboos ; 3.Patients with metastatic disease or recurrent rectal cancer ; 4.Patients with familial adenomatous polyposis ( FAP ), hereditary nonpolyposis colorectal cancer ( HNPCC ), active Crohn 's disease or active ulcerative colitis ; 5.Patients with other malignant tumors within 5 years before enrollment, except for basal cell or squamous cell carcinoma of the skin after radical resection, or cervical carcinoma in situ ; 6.Severe cardiovascular diseases, including unstable angina or myocardial infarction, occurred within 6 months before enrollment ; 7.Subjects who were allergic to the study drug or any of its adjuvants ; 8.Participated in other domestic unapproved or unlisted drug clinical trials within 4 weeks before enrollment and received corresponding experimental drug treatment ; 9.International normalized ratio ( INR ) > 1.5 or activated partial thromboplastin time ( APTT ) > 1.5 × ULN ; 10.Investigators judged clinically significant electrolyte abnormalities ; 11.There was uncontrolled hypertension before enrollment, which was defined as : systolic blood pressure ≥ 140 mmHg and / or diastolic blood pressure ≥ 90 mmHg ; 12.There were poorly controlled diabetes before enrollment ( after regular treatment, fasting glucose concentration ≥ CTCAE grade 2 ) ; 1.3.13.Before enrollment, there are any diseases or states that affect drug absorption, or patients cannot take oral drugs ; 14.Before entering the group, there were gastrointestinal diseases such as gastric and duodenal active ulcers and ulcerative colitis, or other conditions that may cause gastrointestinal bleeding and perforation determined by the researchers ; 15.Severe active bleeding, hemoptysis ( fresh blood > 5 mL within 4 weeks ) or thromboembolic events occurred within 12 months before enrollment ( package ).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
cCR rate | 5 years
  the clinical complete remission rate of short-course radiotherapy followed by sequential fruquintinib combined with PD1 monoantibody therapy for locally advanced rectal cancer.

IPD SHARING:
Plan to Share IPD: No